CLINICAL TRIAL: NCT01401088
Title: Evaluation of Safety and Efficacy of Glaucoma Shunt (Aurolab Artificial Drainage Implant) in Refractory Glaucoma
Acronym: AADI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aurolab (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1PN1011049
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Glaucoma
Keywords: patient with refractory glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Artificial drainage implant (Experimental): Aurolab Artificial Drainage Implant (AADI) on intraocular pressure reduction will be implanted in patients with refractory glaucoma.
  Interventions: Device: Artificial drainage implant

INTERVENTIONS:
Device: Artificial drainage implant — Artificial drainage implant is used for intra ocular pressure reduction in patient with refractory glaucoma
  Other Names: AADI

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Aurolab Artificial Drainage Implant (AADI) on intraocular pressure reduction in patients with refractory glaucoma.

DETAILED DESCRIPTION:
Aurolab Artificial Drainage Implant is a non resistant tube device based on Baerveldt implant. It reduces intra ocular pressure by draining aqueous from anterior chamber into sub-conjunctival space formed around base of the implant. Reduction of intraocular pressure prevents further damage to optic nerve and functional visual field loss in advanced refractory glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Significant optic nerve damage and visual field loss due to glaucoma in eligible eyes
* Eligible eyes is considered at high risk of failure/complication following conventional filtering surgery
* Eyes with uncontrolled glaucoma with prior history of Filtering surgery/Uveitic/ Neovascular/Developmental glaucomas
* IOP≥18 mm of Hg with or without anti glaucoma medications
* If taking glaucoma medications, stable dose for 6 weeks

Exclusion Criteria:

* Age<18 years
* Eyes with uncontrolled glaucoma expected to have favorable post-operative outcome by conventional trabeculectomy
* Corneal abnormalities that would preclude accurate IOP readings
* Uncontrolled systemic diseases
* Endothelial cell count<1800cells/mm
* Any other active ocular disease,(active uveitis, ocular infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Intra Ocular Pressure (IOP) | One year
  Mean Intraocular pressure (IOP) reduction from pre operative IOP

SECONDARY OUTCOMES:
Success rate | one year
  Success rate (defined as Inraocular pressure (IOP) of 5mmHg to 20 mmHg and at least a 20% reduction in IOP without visually devastating complications or additional glaucoma surgery)
Number of patients with adverse events as a measure of safety | one year
  to assess the incidence of post operative adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Prashanth Ranganath, MBBS., MS.,, Principal Investigator — Aravind Eye Hospital, Madurai
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India